CLINICAL TRIAL: NCT05095363
Title: The Palliative Care Planner (PCplanner) for Outpatients Pilot Trial
Brief Title: Palliative Care Planner (PCplanner)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00108264
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-01

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis
Keywords: palliative care; advance care planning
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: The Palliative Care planner (PCplanner) is a mobile app platform that aims to facilitate communication on unmet needs and advance care planning between patients with idiopathic pulmonary fibrosis and their pulmonary clinicians. Participants will be randomized to intervention arm in a 2:1 intervention:control ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCplanner mobile app platform (Experimental): Participants who are randomized to the intervention arm will complete surveys at 3 timepoints and will be given resources on advance care planning via PCplanner, the mobile app platform. They will receive a telephone call by the study team about a week after enrollment to answer any questions about the resources provided. If needs and questions are not resolved quickly after the clinic visit, then another layer of patient support with a telephone call by a palliative care specialist will be provided to the participant to help develop potential management plans.
  Interventions: Behavioral: PCplanner
- Usual Care (No Intervention): Participants who are randomized to the usual care arm will complete surveys at 3 timepoints and receive usual care by pulmonary clinician.

INTERVENTIONS:
Behavioral: PCplanner — A mobile app platform that will display participant survey results to clinicians to facilitate communication on specific needs as well as provide resources on advance care planning to participants.
  Arms: PCplanner mobile app platform

SUMMARY:
The purpose of this research study is to determine the feasibility, acceptability, and evidence for clinical impact of a mobile app-based program called Palliative Care Planner (PCplanner) in addressing needs and promoting advance care planning discussions among patients with idiopathic pulmonary fibrosis and their clinicians.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) affects roughly 6.3 to 76 per 100,000 people of predominantly older adult patients worldwide and is associated with high morbidity and mortality. Patients with such idiopathic pulmonary fibrosis suffer symptom burdens similar to patients with cancer and commonly experience long, costly hospitalizations that often include care in an intensive care unit (ICU). Despite the presence of numerous unmet needs, ILD patients uncommonly receive palliative care because of lack of symptom recognition, supports to provide advanced care planning (ACP) and symptom control, and processes to promote collaboration between primary teams and palliative care specialists to deliver the appropriate level of care. To address this important clinical gap, we propose adapting our existing needs-targeted PCplanner (Palliative Care planner) mobile app platform to the outpatient setting. PCplanner Outpatient will allow patients to report their needs, provide video content to stimulate knowledge of and discussion about more advanced care planning, and assist primary physicians in recognizing the optimal timing of specialist palliative care referral.

ELIGIBILITY:
Inclusion Criteria:

* Patient has diagnosis of idiopathic pulmonary fibrosis
* Patient has GAP (gender, age, physiology) index score ≥ 4
* Patient is established in interstitial lung disease clinic (i.e., has had at least 1 previous clinic visit)

Exclusion Criteria:

* Patient lacks fluency in English sufficient to complete study surveys
* Patient is already seeing palliative care or enrolled in hospice
* NEST score <10 at baseline T1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | Up to 16 weeks
  Number of participants who stated intervention was easy to use as measured by patient survey.
Acceptability of intervention | Up to 16 weeks
  Number of participants who stated they were satisfied with the intervention as measured by patient survey.
Completion of intervention | Up to 16 weeks
  Number of participants who completed all three surveys and intervention telephone visits.
Change in Needs; Existential concerns; Symptoms; and Therapeutic interaction (NEST) scale | Baseline to week 8
  Scale ranges from 0 to 130 with lower score indicates less unmet needs and higher score indicates more unmet needs on issues such as communication, symptoms, social support, and financial stress.
Documentation of advance care planning in electronic health record | Up to 16 weeks
  Includes all or any of the following: code status, healthcare power of attorney, advance directive

SECONDARY OUTCOMES:
Change in Needs; Existential concerns; Symptoms; and Therapeutic interaction (NEST) scale | Baseline to week 16
  Scale ranges from 0 to 130 with lower score indicates less unmet needs and higher score indicates more unmet needs on issues such as communication, symptoms, social support, and financial stress.
Change in Patient Health Questionnaire-9 (PHQ-9) score | Baseline to week 8
  Score ranges from 0 to 27 with lower score indicates no or mild depression and higher score indicates more severe depression.
Change in Patient Health Questionnaire-9 (PHQ-9) score | Baseline to week 16
  Score ranges from 0 to 27 with lower score indicates no or mild depression and higher score indicates more severe depression.
Change in General Anxiety Disorder-7 (GAD-7) score | Baseline to week 8
  Score ranges from 0 to 21 with lower score indicates no or mild anxiety and higher score indicates more severe generalized anxiety.
Change in General Anxiety Disorder-7 (GAD-7) score | Baseline to week 16
  Score ranges from 0 to 21 with lower score indicates no or mild anxiety and higher score indicates more severe generalized anxiety.
Change in Patient Health Questionnaire-10 (PHQ-10) score | Baseline to week 8
  Scores range from 0 to 20 with lower score indicates less bothersome symptoms and higher score indicates more bothersome symptoms.
Change in Patient Health Questionnaire-10 (PHQ-10) score | Baseline to week 16
  Scores range from 0 to 20 with lower score indicates less bothersome symptoms and higher score indicates more bothersome symptoms.
Change in EuroQol - 5 Dimension (EQ-5D) score | Baseline to week 8
  Scores generally range from 0 (poor quality of life) to 1 (best quality of life possible)
Change in EuroQol - 5 Dimension (EQ-5D) score | Baseline to week 16
  Scores generally range from 0 (poor quality of life) to 1 (best quality of life possible)
Change in Quality of Life Visual Analogue Scale (QOL VAS) | Baseline to week 8
  Scores range from 0 to 100 with lower score indicates worse imaginable quality of life and higher score indicates better imaginable quality of life.
Change in Quality of Life Visual Analogue Scale (QOL VAS) | Baseline to week 16
  Scores range from 0 to 100 with lower score indicates worse imaginable quality of life and higher score indicates better imaginable quality of life.
Change in Therapeutic Alliance score | Baseline to week 8
  Score ranges from 16 to 64 with lower score indicates lower perceived alliance between patient and their provider and higher score indicates better therapeutic alliance.
Change in Therapeutic Alliance score | Baseline to week 16
  Score ranges from 16 to 64 with lower score indicates lower perceived alliance between patient and their provider and higher score indicates better therapeutic alliance.

OTHER OUTCOMES:
Number of hospitalizations during study | Up to 16 weeks
  Admission to a hospital abstracted from electronic health record
Referral to palliative care specialist during study | Up to 16 weeks
  Referral to palliative care specialist during study abstracted from electronic health record
Referral to hospice during study | Up to 16 weeks
  Referral to inpatient or home hospice during study abstracted from electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cox, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olson A, Hartmann N, Patnaik P, Wallace L, Schlenker-Herceg R, Nasser M, Richeldi L, Hoffmann-Vold AM, Cottin V. Estimation of the Prevalence of Progressive Fibrosing Interstitial Lung Diseases: Systematic Literature Review and Data from a Physician Survey. Adv Ther. 2021 Feb;38(2):854-867. doi: 10.1007/s12325-020-01578-6. Epub 2020 Dec 14. PMID 33315170
- [Background] Moens K, Higginson IJ, Harding R; EURO IMPACT. Are there differences in the prevalence of palliative care-related problems in people living with advanced cancer and eight non-cancer conditions? A systematic review. J Pain Symptom Manage. 2014 Oct;48(4):660-77. doi: 10.1016/j.jpainsymman.2013.11.009. Epub 2014 May 5. PMID 24801658
- [Background] Gore JM, Brophy CJ, Greenstone MA. How well do we care for patients with end stage chronic obstructive pulmonary disease (COPD)? A comparison of palliative care and quality of life in COPD and lung cancer. Thorax. 2000 Dec;55(12):1000-6. doi: 10.1136/thorax.55.12.1000. PMID 11083884
- [Background] Au DH, Udris EM, Fihn SD, McDonell MB, Curtis JR. Differences in health care utilization at the end of life among patients with chronic obstructive pulmonary disease and patients with lung cancer. Arch Intern Med. 2006 Feb 13;166(3):326-31. doi: 10.1001/archinte.166.3.326. PMID 16476873
- [Background] Bausewein C, Booth S, Gysels M, Kuhnbach R, Haberland B, Higginson IJ. Understanding breathlessness: cross-sectional comparison of symptom burden and palliative care needs in chronic obstructive pulmonary disease and cancer. J Palliat Med. 2010 Sep;13(9):1109-18. doi: 10.1089/jpm.2010.0068. PMID 20836635
- [Background] Bajwah S, Higginson IJ, Ross JR, Wells AU, Birring SS, Patel A, Riley J. Specialist palliative care is more than drugs: a retrospective study of ILD patients. Lung. 2012 Apr;190(2):215-20. doi: 10.1007/s00408-011-9355-7. Epub 2012 Jan 5. PMID 22218887
- [Background] Rabow MW, Dibble SL, Pantilat SZ, McPhee SJ. The comprehensive care team: a controlled trial of outpatient palliative medicine consultation. Arch Intern Med. 2004 Jan 12;164(1):83-91. doi: 10.1001/archinte.164.1.83. PMID 14718327
- [Background] Higginson IJ, Bausewein C, Reilly CC, Gao W, Gysels M, Dzingina M, McCrone P, Booth S, Jolley CJ, Moxham J. An integrated palliative and respiratory care service for patients with advanced disease and refractory breathlessness: a randomised controlled trial. Lancet Respir Med. 2014 Dec;2(12):979-87. doi: 10.1016/S2213-2600(14)70226-7. Epub 2014 Oct 29. PMID 25465642
- [Background] Ley B, Ryerson CJ, Vittinghoff E, Ryu JH, Tomassetti S, Lee JS, Poletti V, Buccioli M, Elicker BM, Jones KD, King TE Jr, Collard HR. A multidimensional index and staging system for idiopathic pulmonary fibrosis. Ann Intern Med. 2012 May 15;156(10):684-91. doi: 10.7326/0003-4819-156-10-201205150-00004. PMID 22586007
- [Background] Ryerson CJ, Vittinghoff E, Ley B, Lee JS, Mooney JJ, Jones KD, Elicker BM, Wolters PJ, Koth LL, King TE Jr, Collard HR. Predicting survival across chronic interstitial lung disease: the ILD-GAP model. Chest. 2014 Apr;145(4):723-728. doi: 10.1378/chest.13-1474. PMID 24114524
- [Derived] Gu J, Wang P, Chow SC, Dempsey K, Bermejo S, Swaminathan A, Soskis A, Fried J, Kloefkorn C, Jones C, Cox CE. An App Platform-Facilitated Collaborative Palliative Care Intervention for Outpatients With Interstitial Lung Disease: A Pilot Randomized Trial. Am J Hosp Palliat Care. 2025 Jul;42(7):653-660. doi: 10.1177/10499091241275966. Epub 2024 Aug 19. PMID 39158903